CLINICAL TRIAL: NCT02324790
Title: A Multicenter Pilot Study on the Indications of Negative Pressure Sleep Therapy System for the Treatment of Obstructive Sleep Apnea (OSA)
Brief Title: Pilot Study of Negative Pressure Sleep Therapy System to Treat Obstructive Sleep Apnea
Status: Terminated | Phase: Not Applicable | Type: Interventional
Sponsor: Somnics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CSP-1401-CIP
Record Dates: First submitted 2014-12-11; First posted 2014-12-24 (Estimated); Last update posted 2018-03-19 (Actual); Status verified 2018-03

CONDITIONS: Obstructive Sleep Apnea
Keywords: OSA, Oral Pressure Therapy (OPT)
MeSH Terms: conditions — Sleep Apnea, Obstructive

STUDY DESIGN:
Masking Description: evaluator blind
Oversight: Data Monitoring Committee: No

ARMS (1):
- Treatment (Experimental): Treated with iNAP® Sleep Therapy System on the treatment PSG night.
  Interventions: Device: iNAP® Sleep Therapy System

INTERVENTIONS:
Device: iNAP® Sleep Therapy System — The iNAP® Sleep Therapy System provides pressure gradient within the oral cavity to pull the tongue toward upper palate and the soft palate forward, which aims to maintain better upper airway patency near the pharynx to prevent sleep-disordered breathing.
  Other Names: Negative Pressre Sleep Therapy System; iNAP®

SUMMARY:
This is a pilot study to investigate the efficacy and safety of the Negative Pressure Sleep Therapy System for the treatment of obstructive sleep apnea.

DETAILED DESCRIPTION:
This is an open-lable, single-arm, evaluator-blind and prospective study aimed to evaluate the feasibility of the Negative Pressure Sleep Therapy System for the treatment of obstructive sleep apnea.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of OSA, based on AHI 10~60 (as assessed per baseline PSG).
* Subject understands the study protocol and is willing and able to comply with study requirements and sign the informed consent form.
* BMI ≦ 28.

Exclusion Criteria:

* Poor nasal patency as evidenced by the inability to breathe through the nose with the mouth closed.
* Oral cavity infection or any other oral or dental condition or problem that would limit subject use of the device. (e.g. dentures, loose tooth/teeth, temporomandibular joint (TMJ) conditions, or any oral or dental condition that the Investigator believes could be exacerbated by the Sleep Therapy System.
* History of any OSA surgical treatment including uvulopalatopharyngoplasty surgery (UPPP), maxillomandibular advancement surgery (MMA), radio frequency (RF) ablation treatment, palatal stent devices, etc.
* History of allergic reaction to silicone.
* Any concomitant diagnosed or suspected sleep or chronic neurological disorders, other than OSA, including insomnia, and central sleep apnea.
* Currently working nights, rotating night shifts, planned travel across four or more time zones required during study period, or within two weeks prior to study enrollment, or sleep schedule not compatible with sleep lab practices.
* Current use of medication or other treatment which, in the investigator's opinion, may pose additional risk to the subject or confound the results of the study.
* Potential sleep apnea complications that, in the opinion of the investigator, may affect the health or safety of the participant, including: low blood oxygen, recent near-miss or prior automobile accident due to sleepiness, reported history of severe cardiovascular disease (including New York Heart Association (NYHA) class III or IV heart failure, CAD with angina or myocardial infarction (MI)/stroke in past 6 months, uncontrolled hypertension or hypotension, cardiac arrhythmias), reported respiratory disorders, or use of medication or other treatment which may pose additional risk to the subject or confound the results of the study.
* Female subjects who are pregnant or intend to become pregnant during the study period.

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2014-12; Primary Completion 2016-01-13 (Actual); Study Completion 2016-01-13 (Actual)

PRIMARY OUTCOMES:
Change from baseline of Apnea-Hypopnea Index (AHI) | One treatment night
  The study was terminated. No enough samples for statistical analysis.

SECONDARY OUTCOMES:
Change from baseline of obstructive apnea reduction | One treatment night
  The study was terminated. No enough samples for statistical analysis.
Change from baseline of oxygen desaturation index (ODI) | One treatment night
  The study was terminated. No enough samples for statistical analysis.
Adverse event (AE)/ serious adverse event (SAE) rate and type | From informed consent form obtained to the end of study, average of 4 weeks
  During the entire study period, a total of only 9 events were reported by 8 patients.

CONTACTS AND LOCATIONS:
Overall Officials: C.M. Lin, M.D., Principal Investigator — Shin Kong Wu Ho-Su Memorial Hospital
Locations (4):
- Taiwan (4):
  - Mackay Memorial Hospital, Hsinchu, Hsinchu
  - China Medical University Hospital, Taichung
  - Shin Kong Wu Ho-Su Memorial Hospital, Taipei
  - Taipei Veterans General Hospital, Taipei